CLINICAL TRIAL: NCT06052423
Title: ARTEMIS-007: A Phase 2 Study to Evaluate Efficacy and Safety of HS-20093 in Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: ARTEMIS-007: HS-20093 in Patients With Extensive Stage Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Research and development strategy adjustment.
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-20093-206
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Extensive Stage Small Cell Lung Cancer (ES-SCLC)
Keywords: Extensive Stage Small Cell Lung Cancer; B7-H3; antibody-drug conjugate (ADC); HS-20093

STUDY DESIGN:
Intervention Model Description: Single Arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-20093 (Experimental): All subjects will receive HS-20093 at 10mg/kg
  Interventions: Drug: HS-20093

INTERVENTIONS:
Drug: HS-20093 — HS-20093 is a fully humanized IgG1 antibody-drug conjugate (ADC) which specifically binds to B7-H3, a target wildly expressed on solid tumor cells.

SUMMARY:
This is a phase 2,open-label, multi-center study to evaluate the efficacy, safety, pharmacokinetics (PK) and immunogenicity of HS-20093 as a monotherapy in patients with small cell lung cancer(SCLC).

DETAILED DESCRIPTION:
Intravenous (IV) administration of HS-20093 Q3W; Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. At least age of 18 years at screening.
2. Pathologically diagnosed as ES-SCLC; no prior systemic therapy for ES-SCLC.
3. At least one measurable lesion according to RECIST 1.1.
4. Agree to provide fresh or archival tumor tissue and peripheral blood samples.
5. ECOG PS of 0~1.
6. Life expectancy >= 12 weeks.
7. Men or women should be using adequate contraceptive measures throughout the study.
8. Females subjects must not be pregnant at screening or have evidence of non-childbearing potential.
9. Signed and dated Informed Consent Form.

Exclusion Criteria:

Treatment with any of the following:

1. Previous or current treatment with B7-H3 targeted therapy
2. Radiotherapy with a limited field of radiation for palliation within 2 weeks, or patients received more than 30% of the bone marrow irradiation, or large-scale radiotherapy within 4 weeks prior to the first scheduled dose of HS-20093.
3. Pleural or peritoneal effusion or pericardial effusion requiring clinical intervention.
4. Major surgery within 4 weeks prior to the first dose of HS-20093.
5. Treatment with drugs that are predominantly CYP3A4 strong inhibitors or inducers or sensitive substrates of CYP3A4 with a narrow therapeutic range within 7 days of the first dose of study drug; or requiring treatment with these drugs during the study.
6. Currently receiving drugs known to prolong QT interval or may cause torsade de pointe; or requiring treatment with these drugs during the study.

   2. Spinal cord compression or brain metastases. 3. CNS metastases with symptomatic or active progression. 4. Patients with tumor invasion of surrounding vital organs and blood vessels, at risk of esophagotracheal or esophagopleural fistula.

   5. Any unresolved toxicities from prior therapy greater than Grade 2 according to CTCAE 5.0.

   6. History of other primary malignancies. 7. Inadequate bone marrow reserve or organ dysfunction 8. Evidence of cardiovascular risk. 9. Severe, uncontrolled or active cardiovascular diseases. 10. Diabetes ketoacidosis or hyperglycemia hypertonic occurring within 6 months before the first dose of the study drug, or the glycosylated hemoglobin value ≥ 7.5% in the screening period.

   11. Severe or poorly controlled hypertension. 12. Bleeding symptoms with apparent clinical significance or obvious bleeding tendency within 1 month prior to the first dose of HS-20093 13. Serious arteriovenous thrombosis events occurred within 3 months before the first dose.

   14. Severe infections occurred within 4 weeks before the first dose. 15. Patients who have received continuous glucocorticoid treatment for more than 30 days within 30 days before the first dose, or need long-term (≥ 30 days) steroid treatment, or who have other acquired and congenital immunodeficiency diseases, or have a history of organ transplantation.

   16. The presence of active infectious diseases has been known before the first dose such as hepatitis B, hepatitis C, tuberculosis, syphilis, or human immunodeficiency virus HIV infection, etc.

   17. Hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh Grade B or more severe cirrhosis.

   18. Other moderate or severe lung diseases. 19. Previous history of serious neurological or mental disorders. 20. Women who are breastfeeding or pregnant or planned to be pregnant during the study period.

   21. Vaccination or hypersensitivity of any level within 4 weeks prior to the first dose of HS-20093 22. History of severe hypersensitivity reaction, severe infusion reaction or allergy to recombinant human or mouse derived proteins.

   23. Hypersensitivity to any ingredient of HS-20093. 24. Unlikely to comply with study procedures, restrictions, and requirements in the opinion of the investigator 25. Any disease or condition that, in the opinion of the investigator, would compromise subject safety or interfere with study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) determined by investigators according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | From the first dose up to disease progression or withdrawal from study, which ever came first, assessed up to 18 months
  ORR was defined as the percentage of participants who achieved a best overall response (BOR) of confirmed Complete Response (CR) or Partial Response (PR), assessed by investigators based on RECIST version 1.1[Confirmed CR/PR assessment require at least one repeat (≥4 weeks)]

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) | From the first dose through 90 days post end of treatment
  AE assessed by investigator exclusively related to subject's underlying disease or medical condition [graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0]. Any untoward medical occurrence in a clinical study participant, whether or not considered related to the medicinal product. Incidence and severity of AEs are assessed according to vital signs, laboratory variables, physical examination, electrocardiogram, etc.
Observed maximum plasma concentration (Cmax) of HS-20093 | From pre-dose to 14 days after the first dose on Cycle 1 (each cycle is 21 days)
  Cmax will be obtained following administration of the first dose of HS-20093 during the first cycle
Time to reach maximum plasma concentration (Tmax) of HS-20093 following the first dose in participants with advanced solid tumor | From pre-dose to 14 days after the first dose on Cycle 1 (each cycle is 21 days)
  Tmax will be obtained following administration of the first dose of HS-20093 during the first cycle
Terminal half-life (T1/2) of HS-20093 following IV dose in participants with advanced solid tumor | From pre-dose to 14 days after the first dose on Cycle 1 (each cycle is 21 days)
  Apparent terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by λz
Area under plasma concentration versus time curve from zero to last sampling time (AUC0-t) following the first dose of HS-20093 | From pre-dose to 14 days after the first dose on Cycle 1 (each cycle is 21 days)
  Area under the plasma concentration versus time curve from time zero to the last sampling time when the concentration was no less than the lower limit of quantification (LLQ). AUC0-t was calculated according to the mixed log-linear trapezoidal rule
Percentage of participants with antibodies to HS-20093 in serum | From pre-dose to 90 days post end of treatment
  Serum samples were collected for the determination of anti-drug antibody (ADA) at designated time points
Disease control rate (DCR) determined by investigators according to RECIST 1.1 | From the first dose up to disease progression or withdrawal from study, whichever came first, assessed up to 18 months
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline. DCR was evaluated by the number of participants with best overall response of CR, PR and stable disease (SD) [Confirmed CR/PR assessment require at least one repeat (≥4 weeks); SD shall be assessed at least 5 weeks after the first dose]
Duration of response (DoR) determined by investigators according to RECIST 1.1 | From the first dose up to disease progression or withdrawal from study, whichever came first, assessed up to 18 months
  DoR was defined as the period from the first occurrence of CR or PR to progressive disease (PD) or death from any cause. If no PD or death after CR/PR, the cut-off date of progression-free survival (PFS) would be used [Confirmed CR/PR assessment require at least one repeat (≥4 weeks)]
Progression-free survival (PFS) determined by investigators according to RECIST 1.1 | From the first dose or random assignment up to disease progression or withdrawal from study, whichever came first, assessed up to 18 months
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline. PFS was defined as the time from first dose or random assignment (if any) to PD or death from any cause
Overall survival (OS) | From the first dose or random assignment up to death or withdrawal from study, whichever came first, assessed up to 18 months
  OS was defined as the time from the first dose or random assignment (if any) to death from any cause